CLINICAL TRIAL: NCT01175070
Title: A Phase IV OpenLabelled Prospective Pilot Study of Intravitreal Macugen (Pegaptanib) for Ischaemic Diabetic Macular Oedema (MIDME Study)
Brief Title: Intravitreal Macugen for Ischaemic Diabetic Macular Oedema
Acronym: MIDME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIDME 001 PID 6180
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Diabetic Macular Oedema
Keywords: diabetic macular oedema; ischaemia; anti VEGF; pegaptanib; Ischaemic diabetic macular oedema
MeSH Terms: conditions — Ischemia | interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pegaptanib (Experimental): Participants receiving 6-weekly treatment with pegaptanib sodium (Macugen [TM]) for ischaemic diabetic macular oedema over a 30 week period.
  Interventions: Drug: Intravitreal injection of pegaptanib sodium

INTERVENTIONS:
Drug: Intravitreal injection of pegaptanib sodium — Eligible participants with ischaemic diabetic macular oedema will receive an intravitreal injection of pegaptanib sodium (Macugen [TM]) 0.3mg every 6 weeks over a 30 week period.
  Other Names: Macugen 0.3mg

SUMMARY:
Diabetic macular oedema (DME) is one of the leading causes of blindness in the United Kingdom's working population. It affects the macula, which lies at the centre of the retina, at the back of the eye. Damage to the macula can occur either because the blood supply is reduced (ischaemic DME), or because the blood vessels are leaking excessively (exudative DME).

A chemical called vascular endothelial growth factor (VEGF) may underlie some of the abnormalities seen in DME. Studies have shown that VEGF encourages leakage of fluid from blood vessels and increases the stickiness of white blood cells. When white blood cells are sticky they can attach to blood vessel walls. This may cause small blood vessels to block, and lead to ischaemia.

Laser treatment often helps to stabilise exudative DME, but there is currently no recognised treatment for ischaemic DME. Macugen (pegaptanib), a drug that inactivates VEGF, has been tried and found to be of benefit in treating exudative DME. Since VEGF promotes ischaemia, it is possible that Macugen will also prove to be beneficial for ischaemic DME. This has not been tested before.

A healthy macula is essential for good vision. The innermost area of the macula, the foveal avascular zone (FAZ), is the most important part. The FAZ is enlarged when it is ischaemic. This is a pilot study to assess whether Macugen can reduce the size of the FAZ in ischaemic DME. The investigators will also assess whether it can reduce retinal thickness and improve vision in ischaemic DME. Thirty patients will be involved in the study for thirty weeks each. They will have their eyes examined and receive an injection of Macugen into the eye every 6 weeks. The study is taking place in the Oxford Eye Hospital and is being funded by Pfizer, the company that makes Macugen.

DETAILED DESCRIPTION:
Diabetic macular oedema:

A combination of increasing longevity and increasing obesity is causing a rise in the incidence of diabetes and its associated complications such as diabetic retinopathy. Almost all patients with type 1 diabetes mellitus (DM) develop some signs of retinopathy and approximately 60% of patients with type 2 DM develop diabetic retinopathy. Of those with type 2 DM, diabetic macular oedema (DME) is the most common cause of reduced visual acuity. [1]

DME is one of the leading causes of loss of vision in people of a working age in the developed world. It affects the function of the macula, a key part of the retina which is used for central vision. In DME there are abnormal structural changes in the blood vessel walls which lead to leakage of fluid and proteins from the blood vessels. [2, 3] DME can be classified as ischaemic or exudative, based on the dominant underlying problem. In ischaemic DME, the main problem is a reduction in blood flow to the macula which causes reduced central vision and swelling of the retinal tissues in this area. [4] In exudative DME, excessive leakage of fluid from the blood vessels around the macula results in thickening or swelling of the retina and a resultant reduction in central vision. There is often a combination of ischaemia and exudation.

Vascular endothelial growth factor:

A chemical called vascular endothelial growth factor (VEGF) has been implicated as a potential cause of the abnormalities seen in DME. It has been shown to modulate the growth and pattern of blood vessels, the tone and permeability of their walls, and to cause white blood cells to be drawn to the inner walls of blood vessels. [5, 6] The actual roles played by VEGF are in part dependent on the needs of the tissues in which it is acting. [5] Studies of diseases of the eye that involve the abnormal development of new blood vessels, such as neovascular age-related macular degeneration (AMD) and proliferative diabetic retinopathy (PDR), have demonstrated a central role for VEGF. It has also been implicated in the development of some of the problems associated with central retinal vein occlusion (CRVO) and DME. VEGF exists in a variety of subtypes, called "isoforms", each described by the number of amino acids (the building blocks of proteins) that it contains. The different VEGF isoforms have distinct activities at different sites in the body and its various tissues. [7] This may in part help to explain how VEGF is able to elicit such a variety of functions within blood vessels and beyond. [5]

A role for VEGF inhibitors in the eye:

Macugen [TM] (OSI-Eyetech, Inc. and Pfizer, Inc.), also known as pegaptanib, is a drug which has the ability to block one of the isoforms of VEGF called VEGF(165), leaving the other types of VEGF unaffected [8]. It inhibits the amount of leakage of fluid through blood vessel walls. It has been demonstrated that VEGF(165) alone mediates abnormal new blood vessel development in the eye, and its inactivation by Macugen [TM] inhibits the new vessel development observed in patients with neovascular AMD [8] without affecting normal blood vessel development, which is supported by the VEGF(121) isoform. In addition, animal model studies have shown that injection of Macugen [TM] into the fluid at the back of the eye ("intravitreal injection") can inhibit or even show signs of reversing the typical damage to the blood vessels that occurs in diabetes. [9] These findings suggest that that intravitreal Macugen [TM] could provide a safe and effective treatment against both the development of abnormal new blood vessels in the eye and diabetes-induced damage to the blood vessels of the retina. [6] They formed the basis for randomized controlled trials examining the efficacy of Macugen [TM] as a therapy for AMD and DME. [8]

Other inhibitors of VEGF or "antiVEGF" drugs exist. These include Avastin [TM] (bevacizumab, Genentech, Inc) and Lucentis [TM] (ranibizumab, Genentech, Inc.) which bind to and inhibit all VEGF isoforms, in contrast to Macugen [TM] which is specific for VEGF(165). To date, Macugen [TM] and Lucentis [TM] have received regulatory approval for the treatment of neovascular AMD. Increasingly antiVEGF drugs are being examined to see if they might play a beneficial role in other ocular conditions.

The generalized leakage of fluid from tiny blood vessels ("capillary hyperpermeability") seen in DME has been described as being somewhat analogous to the leakage or "hyperpermeability" seen from the abnormal blood vessels (choroidal neovascularisation) associated with AMD. [10] Therapeutic effects from blockade of the VEGF(165) isoform previously demonstrated in AMD have been demonstrated in DME. That particular study, detailed below, did not specify the degree of macular ischaemia that these patients had.

Safety and efficacy of Macugen [TM] were assessed in a randomized, sham-controlled, double-masked, Phase 2 trial enrolling 172 diabetic subjects with DME affecting the centre of the fovea. The participants were individuals with a best-corrected visual acuity (BCVA) between 20/50 and 20/320 in the study eye and DME involving the centre of the macula for whom the investigator judged laser photocoagulation (at present the standard treatment for clinically significant exudative DME) could be safely withheld for 16 weeks. Intravitreal injections of Macugen [TM], or a sham injection, were administered at baseline and every six weeks thereafter. At Week 36, 0.3 mg Macugen [TM] was significantly superior to sham injection. The results suggested an overall visual acuity (VA) gain as well as a reduced risk of VA loss in eyes with DME treated with intravitreal Macugen [TM]. The 0.3 mg dose seemed to be the most efficacious dose studied, but due to the relatively small number of participants in the study, the authors were unable to identify statistical differences between the different doses given.

The authors felt that these results were consistent with established and known effects of selective blockade of VEGF(165) bioactivity- decreased leakage from blood vessel walls-and postulated that they suggest an anti-permeability effect at the macula. Most adverse events were transient, mild to moderate in severity, and attributed to the injection and the preparation procedure itself, rather than to the study drug. Macugen [TM] was equally well tolerated systemically, with no apparent increased risk of cardiac, ischaemic or haemorrhagic adverse events. [11] Rates of serious injection-related complications, most notably infection inside the eye (endophthalmitis), were within the range of historical benchmarks of injections into the eye and not associated with severe visual loss. These preliminary findings provide evidence that selective inhibition of VEGF(165) may produce a clinically meaningful and statistically significant benefit in the treatment of DME. Confirmation of these preliminary observations of Macugen [TM] safety, patient tolerance, and significant efficacy across a broad spectrum of patients with DME is required. [10]

There is now a growing body of evidence [12, 13] that suggests that there may be a role for antiVEGF drugs, both selective and unselective, in the treatment of the wide range of ocular conditions caused by the development of abnormal blood vessels, including exudative DME. [14] Results of large, randomised, controlled trials are needed to confirm early safety and efficacy findings from small, open-label prospective studies. Laser photocoagulation treatment, however, remains the current best treatment for clinically significant exudative DME. The primary aim of this type of laser treatment is to try to stabilise vision rather than to improve it. [15] In ischaemic diabetic maculopathy laser treatment is not an option as it would be expected to make vision worse. There is no known effective treatment for ischaemic DME, the natural history of which is of a gradual decline in central vision. Ischaemia is well known to be a major factor in the development and progression of diabetic retinopathy (DR). It may be due in part to the effects of VEGF on the tone of blood vessel walls and narrowing of small blood vessels. Consequently some studies have been done to try to assess the effect of antiVEGF treatment on retinal ischaemia. The results in the literature are conflicting.

VEGF inhibitors and retinal ischaemia:

Neubauer and colleagues [16] showed that the anti-VEGF drug Avastin [TM], which inhibits all isoforms of VEGF, caused a reduction in peripheral retinal ischaemia and an improvement in visual acuity in patients with diabetic retinopathy. They investigated changes in central and peripheral ischaemia after intravitreal injection of Avastin [TM] and were able to demonstrate in a small series of patients with DR that Avastin [TM] treatment improved peripheral ischaemia in the short term. They saw no evidence of increasing ischaemia, as might be feared. Limitations of their study include the small number of patients and short follow-up after only one administration. They believe that the observed reduction of ischaemia makes anti-VEGF therapy a promising approach in the treatment of DR, but further investigations with longer follow-up times are needed.

In contrast, a single case report [17] demonstrated a deterioration in VA with the use of Avastin [TM] for chronic, refractory DME in a 58-year-old woman who had undergone multiple previous treatments including laser photocoagulation and intravitreal triamcinolone (steroid) injections. The authors felt that using Avastin [TM] in this way exacerbated macular ischaemia by disrupting an already fragile perfusion status. It is difficult to attribute the poor outcome fully to the antiVEGF drug, but the report highlights our need to examine the effects of antiVEGF in ischaemic DME more closely.

Chung and colleagues [18] retrospectively analysed the effect of macular ischaemia on the outcome of treatment of DME with Avastin [TM]. They collected data on 59 eyes of 53 consecutive patients and analysed their preoperative imaging tests (fluorescein angiograms) for signs of ischaemia. They then divided the patients into two groups, those with and without signs of ischaemia, in order to assess their outcomes. 3 months after treatment, the group with ischaemia showed a reduction in visual acuity from approximately 20/63 to 20/80, whereas the group without ischaemia showed an improvement in visual acuity from 20/100 to 20/80. Nine of 18 eyes (50%) in the ischaemic group, but only 9 of 41 eyes (21%) in the non-ischaemic group, experienced visual losses of >or=1 line on the ETDRS chart (P = 0.031, Pearson chi-square test). Four eyes (22%) in the ischaemic group, but only 2 eyes (5%) in the non-ischaemic group, lost >or=3 lines (P = 0.042, Pearson chi-square test). Whilst these data show a poorer outcome for patients with macular ischaemia treated with Avastin [TM], compared to those without, they do not show how treatment with Avastin [TM] compares to what would have happened to these patients' vision without any treatment at all. As already discussed the natural history of ischaemic DME is of a decline in visual acuity and there is currently no established treatment option. The investigators would not expect the patients with ischaemic DME to do as well as those without ischaemia as they tend to have much more severe disease than those without ischaemia. In this particular group it appears that the baseline acuity was much poorer in the non-ischaemic group, which gave them more scope for improvement in visual acuity with treatment than the non-ischaemic group which had, on average, better visual acuity, and probably much less oedema, to begin with.

Macugen [TM] for ischaemic DME:

The investigators have chosen to look at Macugen [TM] because of its specificity and generally good safety profile which has now been validated over >4 years. It is possible that a non-selective VEGF inhibitor that blocks all VEGF isoforms could be more deleterious to retinal function over the long term than a more selective VEGF antagonist that could spare several of the smaller soluble VEGF isoforms within the eye. [19] No increased risk of serious systemic adverse events has been shown in any of the major clinical trials of Macugen [TM]. [11] The incidence of ocular adverse events when used for treating AMD is low [20]. As discussed above, Macugen [TM] has been used with benefit in exudative DME but its effectiveness in ischaemic DME, for which there is currently no available treatment, remains unknown.

The investigators plan to use Macugen [TM] to treat 30 patients with ischaemic DME. The investigators will diagnose macular ischaemia by assessing the size of the foveal avascular zone (FAZ). This is the area at the centre of the macula. It is usually devoid of blood vessels in order to maximise visual clarity. The FAZ may be abnormally enlarged and irregular in patients with diabetes and this is a requirement for the diagnosis of ischaemic DME. Enlargement of the FAZ is thought to be a sign of reduced blood flow, possibly related to the effects of VEGF, and is associated with reduced vision. Macugen [TM] will be given at the standard dose that is used for treating AMD and that which was identified as most effective in the phase 2 study of Macugen [TM] in DME, i.e. 0.3mg. Our primary outcome will be the change in size of the FAZ and secondarily we would like to look for a change in thickness of the retina at the centre of the macula or a change in visual acuity. The investigators hope that this pilot study will clarify whether Macugen [TM] might be able to reverse some of the effects of VEGF(165) and be of benefit for those with ischaemic DME, the more severe end of the DME spectrum.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* DME
* BCVA 20/32 to 20/320 inclusive
* Central OCT thickness > 300 microns
* Enlargement of FAZ (ischaemia or capillary drop out of >30% on FFA)
* Female participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
* Able (in the Investigator's opinion) and willing to comply with all study requirements e.g. attending for tests and treatment every 6 weeks.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Any co-existing ocular disease (with the exception of cataract)
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* Any significant disease or disorder, e.g. recent stroke or myocardial infarction, which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study
* Significant renal impairment, i.e. creatinine clearance < 20mL/min
* Participants who have participated in another research study involving an investigational product in the past 12 weeks
* Laser within 3 months
* Intraocular surgery within 6 months
* Known allergy to pegaptanib (Macugen [TM])
* Known allergy to fluorescein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in size of FAZ at 30 weeks | 30 weeks

SECONDARY OUTCOMES:
Change in central foveal thickness and best corrected visual acuity at 30 weeks. | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Victor Chong, MPhil, MD, FRCSEd, FRCOphth, Principal Investigator — Oxford Eye Hospital
Locations (1):
- Oxford Eye Hospital, Oxford, Oxfordshire, United Kingdom